CLINICAL TRIAL: NCT05177562
Title: Reproductive Endocrinology Oxford Study (RepOx)
Acronym: RepOx
Status: Recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Bayer (Industry); Li Ka Shing Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS302159
Record Dates: First submitted 2021-12-15; First posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, saliva, fat, ovarian tissue, endometrium biopsy, cumulus/granulosa cells, follicular fluid.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- PCOS: No intervention.
  Interventions: Other: No intervention
- PCOS surgery: No intervention
  Interventions: Other: No intervention
- Surgery control: No intervention
  Interventions: Other: No intervention
- IVF PCOS: No intervention
  Interventions: Other: No intervention
- IVF control: No intervention
  Interventions: Other: No intervention
- Investigations, fertility PCOS: No intervention
  Interventions: Other: No intervention
- Investigations, fertility control: No intervention
  Interventions: Other: No intervention
- Pregnancy - gestational diabetes mellitus: No intervention
  Interventions: Other: No intervention
- Pregnancy - Intrahepatic cholestasis of pregnancy: No intervention
  Interventions: Other: No intervention
- Pregnancy - control: No intervention
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There is no intervention in this study

SUMMARY:
This is a prospective observational study that aims to identify the underlying mechanisms of PolyCystic Ovarian Syndrome (PCOS) and associated comorbidities such as subfertility, miscarriage; and pregnancy complications such as gestational diabetes mellitus and Intrahepatic cholestasis of pregnancy (ICP). This will be achieved through cross-sectional observation and laboratory analyses.

DETAILED DESCRIPTION:
Here we propose a comprehensive program to dissect the underlying disease-causing mechanisms of PCOS and associated comorbidities. We will investigate how the different layers of biological information (ranging from DNA variant genotyping, to RNA sequencing and proteomics), and clinical characteristics are correlated with each other and how this affects PCOS in fat tissue derived cells, as well as ovarian tissue and tissue derived cells by using a combination of big data analysis, a range of "-omics" technologies, of both in-house generated and publicly available data, paired with state of the art statistical and bioinformatics analysis. Out of these mechanisms and pathways we will identify druggable targets for proposals for detailed functional follow up with an aim of development of novel therapeutic options for PCOS.

ELIGIBILITY:
Inclusion Criteria:

* ● General Criteria for all groups

  * Participant is willing and able to give informed consent for participation in the study.
  * Female, aged between 16 and 45 years of age. As IVF is not undertaken in women less that 18 years, this group will between 18 and 45 years o

    ● PCOS (Group 1, 2 and 3)
  * Currently under investigation for or having diagnosis of PCOS having displayed one or more of the following: Hyperandrogenism, Ovulation Dysfunction and Polycystic ovaries on ultrasound (known as the Rotterdam criteria)

    ● PCOS Controls (Group 4 and 5)
  * Patients under gynaecological investigation or having assisted reproduction
  * Exhibit no features of PCOS

    ● Miscarriage Group (Group 6)
  * Have had at least two previous miscarriages
  * Recruited at any time after their second menstrual cycle following a miscarriage

    ● Miscarriage Controls (Group 7)
  * Patients will have had zero or no more than one miscarriage and having fertility investigations.

    ● Pregnant GDM (Group 8)
  * Pregnant women at least 28 weeks gestation with :
  * 1) A fasting plasma glucose of 5.1mmol/L or above or
  * 2) A 1 hr plasma glucose of 10mmol/L or
  * 3) A 2-hr plasma glucose level of 8.5mmol/L or above

    ● Pregnant ICP (Group 9)
  * Women at least 28 weeks gestation with :
  * Raised ALT or raised bile acids in the context of pruritus with no rash
  * ALT (>32iu/l) and bile acids (>14micromol/l) Pregnant Control (Group 10)
  * Pregnant women at least 28 weeks gestation with no diagnosis of GDM or ICP

Exclusion Criteria:

* For all groups - The participant may not enter the study if ANY of the following apply.

  * Unable to read, or to understand written or spoken English
  * Currently involved in any Clinical Trial of an Investigational Medicinal Product (CTIMP)
  * Undergoing surgery because of a possible cancer diagnosis
  * Diagnosis of other androgen excess disorders such as Congenital Adrenal Hyperplasia (CAH), Androgen Secreting tumours, Cushing syndrome, or Hyperprolactinemia

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Women with and without OCOS and known associated phenotypes
Sampling Method: Non-Probability Sample
Enrollment: 1175 (Estimated)
Dates: Start 2021-10-21 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Identify the underlying genetic and pathophysiological mechanisms of PCOS and associated phenotypes | one visit
  Questionnaire data, imaging analysis, medical records and sample analysis

SECONDARY OUTCOMES:
To identify novel biomarkers of PCOS and associated comorbidities. | one visit
To identify clinical subgroups of PCOS and associated comorbidities. | one visit
To understand the genetics underlying these conditions and explore the relevant downstream molecular pathways | one visit
To identify novel drug targets, develop models of disease progression and prediction. | one visit

CONTACTS AND LOCATIONS:
Locations (1):
- Nuffield Department Women's and Reproductive Health, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No